CLINICAL TRIAL: NCT02225405
Title: Phase I Study of Induction Cisplatin, Docetaxel, and Nintedanib for Stage IB-IIIA Non-Small Cell Lung Cancers Amenable for Surgical Resection
Brief Title: Cisplatin, Docetaxel, and Nintedanib Before Surgery in Treating Patients With Previously Untreated Stage IB-IIIA Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0844; NCI-2014-02091 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013-0844 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Stage IB Non-Small Cell Lung Carcinoma AJCC v7; Stage II Non-Small Cell Lung Cancer AJCC v7; Stage IIA Non-Small Cell Lung Carcinoma AJCC v7; Stage IIB Non-Small Cell Lung Carcinoma AJCC v7; Stage IIIA Non-Small Cell Lung Cancer AJCC v7
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; Docetaxel; nintedanib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cisplatin, docetaxel, nintedanib) (Experimental): RUN-IN PHASE: Patients receive induction therapy comprising cisplatin IV over 2 hours on day 1, docetaxel IV over 1 hour on day 1, and nintedanib PO BID from day 2 of course 1 to day 7 of course 3. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.
  EXPANSION PHASE: Patients receive single-agent nintedanib PO BID on days 1-28. Patients then receive 3 courses of induction chemotherapy and undergo surgery as above. Treatment continues even if patients experience disease progression, unless treatment is judged to be not in the best interest of the patient by the treating physician.
  Interventions: Drug: Cisplatin; Drug: Docetaxel; Other: Laboratory Biomarker Analysis; Drug: Nintedanib

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Docetaxel — Given IV
  Other Names: Docecad; RP56976; Taxotere; Taxotere Injection Concentrate
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nintedanib — Given PO
  Other Names: BIBF 1120; BIBF-1120; Intedanib; Multitargeted Tyrosine Kinase Inhibitor BIBF 1120; tyrosine kinase inhibitor BIBF 1120; Vargatef

SUMMARY:
This phase I trial studies the side effects and best dose of nintedanib when given together with cisplatin and docetaxel and to see how well they work in treating patients with previously untreated stage IB-IIIA non-small cell lung cancer who are undergoing surgery. Drugs used in chemotherapy, such as cisplatin and docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Nintedanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving cisplatin, docetaxel, and nintedanib before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine safety of nintedanib incorporated to chemotherapy in the induction setting.

II. To determine the major pathologic response rate in patients treated with induction nintedanib and chemotherapy.

SECONDARY OBJECTIVES:

I. Response rates to induction treatment (by Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1).

II. Response rates to priming therapy with nintedanib single agent (by computed tomography [CT] assessment using RECIST version 1.1).

III. Recurrence-free survival. IV. Overall survival. V. Correlations between major pathologic response with recurrence-free and overall survival.

VI. Toxicity (assessed by the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE] version 4).

VII. Peri-operative morbidity and mortality. VIII. Complete resection (R0) rate. IX. Correlations of response assessed by imaging studies with outcomes (both pathologic response to treatment and long-term recurrence-free survival).

X. Correlations of blood- and tissue-based biomarkers with efficacy and toxicity.

OUTLINE: This is a dose-escalation study of nintedanib.

RUN-IN PHASE: Patients receive induction therapy comprising cisplatin intravenously (IV) over 2 hours on day 1, docetaxel IV over 1 hour on day 1, and nintedanib orally (PO) twice daily (BID) from day 2 of course 1 to day 7 of course 3. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo surgery.

EXPANSION PHASE: Patients receive single-agent nintedanib PO BID on days 1-28. Patients then receive 3 courses of induction chemotherapy and undergo surgery as above. Treatment continues even if patients experience disease progression, unless treatment is judged to be not in the best interest of the patient by the treating physician.

After completion of study treatment, patients are followed up within 8 weeks and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed non-small cell lung cancer; patients with a suspected lung cancer are eligible, but pathology must be confirmed prior to initiating treatment on study; neuroendocrine carcinomas are not eligible; carcinomas with neuroendocrine differentiation are eligible
* Stage IB (with a primary tumor >= 4 cm), IIA, IIB, or IIIA (according to American Joint Committee on Cancer [AJCC] 7th edition); patients with stage IIIA must not have more than one mediastinal lymph node station involved by tumor
* All patients must have lymph node evaluation of contralateral stations 2 and/or 4 to exclude N3 disease
* The patient must be a suitable candidate for surgery, in the opinion of the treating physician
* Eastern Cooperative Oncology Group (ECOG) performance status score 0-1
* Signed and dated written informed consent prior to admission to the study in accordance with International Conference on Harmonization of Technical Requirements for Registration of Pharmaceuticals for Human Use (ICH)-Good Clinical Practice (GCP) guidelines and to the local legislation

Exclusion Criteria:

* Prior systemic therapy or radiation therapy for treatment of the current lung cancer
* Known hypersensitivity to the trial drugs or to their excipients
* Centrally located tumors with radiographic evidence (CT or magnetic resonance imaging [MRI]) of local invasion of major blood vessels
* Major injuries within the past 10 days prior to start of study treatment with incomplete wound healing
* History of clinically significant hemorrhagic or thromboembolic event in the past 6 months
* Known inherited predisposition to bleeding or thrombosis
* Significant cardiovascular diseases (i.e. uncontrolled hypertension, unstable angina, history of infarction within the past 12 months prior to start of study treatment, congestive heart failure > New York Heart Association [NYHA] II, serious cardiac arrhythmia, pericardial effusion)
* Creatinine > 1.5 x the upper limit of normal; patients with creatinine > 1.5 x the upper limit of normal who have creatinine clearance >= 60 cc/min (calculated using the Cockcroft and Gault equation) are eligible
* Total bilirubin > institutional upper limit of normal or
* Aspartate aminotransferase (AST) > 1.5 x institutional upper limit of normal
* International normalized ratio (INR) > 2
* Prothrombin time (PT) and partial thromboplastin time (PTT) > 50% of deviation of institutional upper limit of normal (ULN)
* Absolute neutrophil count (ANC) < 1500/ml, and/or
* Platelets < 100000/ml
* Prior malignancy requiring systemic therapy or radiation therapy within 1 year of randomization
* Active serious infections in particular if requiring systemic antibiotic or antimicrobial therapy
* Known disease or history of active or chronic hepatitis C and/or B infection
* Gastrointestinal disorders or abnormalities that would interfere with absorption of the study drug
* Serious illness or concomitant non-oncological disease such as neurologic, psychiatric, infectious disease or laboratory abnormality that may increase the risk associated with study participation or study drug administration and in the judgment of the investigator would make the patient inappropriate for entry into the study
* Patients who are sexually active, with preserved reproductive capacity, and unwilling to use a medically acceptable method of contraception (e.g. such as implants, injectables, combined oral contraceptives, some intrauterine devices or vasectomized partner for participating females, condoms for participating males) during the trial and for at least three months after end of active therapy
* Pregnancy or breast feeding
* Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-04-03 (Actual); Primary Completion 2024-05-06 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) of nintedanib | 21 days
  Will be determined according to incidence of dose-limiting toxicity as graded according to National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.
Major pathologic response rate, defined as less than or equal to 10% viable tumor cells in the resected specimen using the methods described by Pataer | Up to 5 years
  Multivariate analysis will be used to explore the role of biomarkers in predicting pathologic response to treatment, in an exploratory way.

SECONDARY OUTCOMES:
Change in tumor size (Expansion phase) | Baseline to 4 weeks
  Will be assessed by computed tomography (CT) after single-agent nintedanib.
Response rate after single-agent nintedanib (Expansion phase) | Up to 4 weeks
  Will be evaluated by Response Evaluation Criteria in Solid Tumors (RECIST).

CONTACTS AND LOCATIONS:
Overall Officials: Tina Cascone, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org